CLINICAL TRIAL: NCT00612274
Title: Pilot Study of Sirolimus, Tacrolimus and Short Course Methotrexate for Prevention of Acute Graft Versus Host Disease in Recipients of Mismatched Unrelated Donor Allogeneic Stem Cell Transplantation
Brief Title: Sirolimus, Tacrolimus and Short Course Methotrexate for Prevention of Acute GVHD in Recipients of Mismatched Unrelated Donor Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0703002455
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Stem Cell Transplantation
Keywords: allogeneic
MeSH Terms: interventions — Tacrolimus; Sirolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): sirolimus, tacrolimus and short course methotrexate
  Interventions: Drug: tacrolimus; Drug: Sirolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: tacrolimus — Tacrolimus will be administered at a dose of .02mg/kg/d IVCI beginning day -3 until able to take oral medicines reliably. Blood levels will be maintained at 5-10 ng/ml. The oral dose will be 4 times the IV dose. Tacrolimus will be converted to oral dosing prior to hospital discharge. Tacrolimus will be continued until 4 months post transplant (day +120) unless toxicity, refractory GVHD or the development of disease recurrence mandate discontinuation of the drug.
  Other Names: FK506; Prograf(TM)
Drug: Sirolimus — Sirolimus will be administered as a 12 mg oral loading dose on day -3 followed by 4mg daily. Sirolimus levels will be obtained on day +0 and then at least twice weekly to maintain a trough serum level of 3-12 ng/ml. Sirolimus will be continued until 5 months post transplant (day +150) unless toxicity, refractory GVHD or the development of disease recurrence mandate discontinuation of the drug.
  Other Names: Rapamune
Drug: Methotrexate — Methotrexate, dose #1 will be administered on day +1 post transplantation, as an IV bolus, provided at least 24 hours have elapsed following infusion of donor stem cells at a dose of 10mg/m2. Dose #2 of Methotrexate will be administered 48 hours later, as IV bolus on day +3 at a dose of 5mg/m2.

SUMMARY:
The primary objective of this trial is to study the safety and efficacy of a novel regimen of sirolimus, tacrolimus and methotrexate as prophylaxis against acute graft versus host disease (GVHD) in recipients of mismatched unrelated donor stem cell grafts. Methotrexate is administered in a low dose format of 5mg/m2 on days +1,3 and 6 only.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an identified 8/10 or 9/10 matched unrelated donor identified following a formal search with confirmatory typing through the national marrow donor program as the best available donor. No matched sibling or fully matched unrelated donor has been identified. HLA typing of donor and recipient will be performed by high resolution molecular typing at HLA A, B, C and DRB1/DQ loci. Patients whose best available donor is matched at 8/10 loci must have at least one of the mismatches at the DQ locus. (no more than one mismatch at HLA A,B,C,DR allowed).
* Candidates for this trial will meet the following criteria:

  1. Adequate organ function for conditioning type:

     For patients receiving ablative conditioning
     * Left Ventricular ejection fraction >45%
     * DLCO >50%
     * Creatinine <1.5
     * Hepatic enzymes <3x upper limit of normal.
     * KPS >70%

     For patients receiving non-ablative conditioning:
     * KPS >70%
  2. Patients with the following diseases will be considered eligible:

     * AML in first remission with high risk features (poor risk cytogenetic abnormalities9, persistent elevated blast count on day +15 or recovery marrow after induction therapy).
     * AML beyond first remission
     * ALL in first remission with high risk features (ph+, t4:11)
     * ALL beyond first remission
     * High risk Myelodysplasia (RAEB-II, RAEB-I with poor-risk cytogenetics)
     * Recurrent Aggressive Non-Hodgkins or Hodgkins lymphoma (indolent histologies excluded) who have failed autologous transplant or have had inadequate response to salvage therapy.
     * CML with transformation
     * CLL with transformation or Fludarabine failure.
     * Severe aplastic anemia with recurrence or failure after immunosuppressive therapy.

Exclusion Criteria:

* Prior allogeneic transplantation
* Active CNS leukemia.
* Female patients who are pregnant or breast feeding
* Karnofsky performance status <70%.
* Active viral, bacterial or fungal infection.
* Patients seropositive for HIV -1,2; HTLV -1,2 (due to the additional immunodeficiency induced by transplantation and immunosuppressive therapy) Requirement for antifungal prophylaxis with Voriconazole for the first 30 days is prohibited.
* Patients not providing informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety/Efficacy of a novel regimen of sirolimus, tacrolimus and methotrexate | Upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Seropian, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States